CLINICAL TRIAL: NCT02384980
Title: Saving Life and Limb: Functional Electrical Stimulation for the Elderly With Peripheral Artery Disease
Brief Title: Saving Life and Limb: FES for the Elderly With PAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MultiCare Health System Research Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14.12; 1R21AG048001-01 (NIH)
Record Dates: First submitted 2014-11-10; First posted 2015-03-10 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Peripheral Arterial Disease
Keywords: Intermittent Claudication; Functional Electrical Stimulation
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walk Group (No Intervention): This group of patients are part of the walk group. They will be encouraged to walk and will receive standard care, defined as conservative (non-surgical) management of signs and symptoms, including prescriptive medications to improve circulation and manage pain, determined by their attending physician on a case by case basis.
- FES + Walk Group (Experimental): This group of patients will participate in Functional Electrical Stimulation (FES) and exercise. This group will receive functional electrical stimulation as an intervention. The FES device will stimulate (activate) the calf and shin leg muscles of both legs while the patient is walking. This group will also receive standard care, defined as conservative (non-surgical) management of signs and symptoms, including prescriptive medications to improve circulation and manage pain, determined by their attending physician on a case by case basis.
  Interventions: Device: FES (Gait MyoElectric Stimulator)

INTERVENTIONS:
Device: FES (Gait MyoElectric Stimulator) — Functional Electrical Stimulation (FES) will be tested in a group of peripheral arterial disease patients using the Gait MyoElectric Stimulator. The FES device will be applied to the calf and shin muscles on both of the patients legs.
  Arms: FES + Walk Group

SUMMARY:
This study will take the first step to improve public health for millions of Americans with Peripheral Arterial Disease who have extreme difficulty walking due to leg pain. The investigators will assess a proof of concept, home administered, functional electrical stimulation (FES) system to resolve pain, improve walking, and enhance quality of life.

DETAILED DESCRIPTION:
This study will evaluate an innovative approach to reduce the debilitating symptoms of peripheral arterial disease (PAD) and ischemic pain during walking (intermittent claudication) by using a new Functional Electrical Stimulation (FES) system. The investigators hypothesize that combining the FES and walking one hour/day (FES+Walk) will significantly reduce pain during walking, improve locomotion, and enhance quality of life when compared to walking one hour/day (Walk) alone after 8 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients who:

1. Are ambulatory, community dwelling adults with evidence of PAD including ankle/brachial index ABI=0.4-0.9
2. Have symptom severity of Fontaine stage II-III
3. Have a score of 24 or higher on the Folstein Mini Mental test
4. Have visible muscle contraction of the plantar flexor (PF) and dorsiflexor (DF) muscles using FES

Exclusion Criteria:

Patients who:

1. Have an electronic implanted stimulator such as pacemaker, defibrillator, deep brain stimulator, spinal cord stimulator
2. Are pregnant
3. Cannot walk without a walker or require human assistance to walk,
4. Present with arthritis or neurological damage resulting in paresis or paralysis of the lower extremity
5. Have skin lesion(s) on the legs where the FES is placed

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from initial assessment, baseline, end of intervention and final assessment using the Perceived Pain Intensity Scale | Initial, baseline assessment, assessment at the end of 8 weeks intervention and final assessment at 16 weeks (8 weeks post-intervention)
  We will measure the changes in pain scores from baseline to end of intervention and end of post-intervention
Change from initial assessment, baseline, end of intervention and final assessment using the 6 Minute Walk Test | Initial, baseline assessment, assessment at the end of 8 weeks intervention, and final assessment at 16 weeks (8 weeks post- intervention)
  We will measure the changes in distance walked during the 6 minute walk test
Change from initial assessment, baseline, end of intervention and final assessment using the Peripheral Artery Disease Quality of Life Questionnaire | Initial, baseline assessment, assessment at the end of 8 weeks intervention and final assessment at 16 weeks (8 weeks post- intervention)
  We will record and measure the changes in questionnaire scores from baseline to end of intervention and end of post-intervention

SECONDARY OUTCOMES:
Change from initial assessment, baseline, end of intervention and final assessment using the Timed-Up-and-Go test | Initial, baseline assessment, assessment at the end of 8 weeks intervention and final assessment at 16 weeks (8 weeks post- intervention)
  We will measure the time (seconds) to complete the test from baseline to end of intervention and end of post-intervention
Change from initial assessment, baseline, end of intervention and final assessment using the Intermittent Claudication Questionnaire (ICQ) | Initial, baseline assessment, assessment at the end of 8 weeks intervention and final assessment at 16 weeks (8 weeks post- intervention)
  We will record and measure the questionnaire score from baseline to end of intervention and end of post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: David G. Embrey, PT, PhD, Principal Investigator — Principal Investigator
Locations (1):
- MultiCare Health System, Tacoma, Washington, United States

REFERENCES:
- [Derived] Embrey DG, Alon G, Brandsma BA, Vladimir F, Silva A, Pflugeisen BM, Amoroso PJ. Functional electrical stimulation improves quality of life by reducing intermittent claudication. Int J Cardiol. 2017 Sep 15;243:454-459. doi: 10.1016/j.ijcard.2017.05.097. Epub 2017 Jun 2. PMID 28595744
- See also: An introductory article about this NIH funded study and benefits of functional electrical stimulation — http://www.multicare.org/news/multicare-researcher-wins-nih-grant/